CLINICAL TRIAL: NCT02564952
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Study to Investigate Possible Drug-drug Interactions Between Clobazam and Cannabidiol (GWP42003-P)
Brief Title: An Open-label Extension Study to Investigate Possible Drug-drug Interactions Between Clobazam and Cannabidiol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GWEP1428 Open-Label Extension; 2014-002942-33 (EudraCT Number)
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy
Keywords: Cannabidiol (CBD); GWP42003-P; Clobazam; Epidiolex
MeSH Terms: conditions — Epilepsy | interventions — Cannabidiol; Clobazam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GWP42003-P (Experimental): Participants who transferred from the DB phase (NCT02565108) to the OLE (still blinded at that stage) tapered off their GWP42003-P or placebo treatment by reducing their maintenance dose by 10% per day and concomitantly titrating GWP42003-P to 20 mg/kg/day initially for the OLE; doses could then be adjusted up or down, dependent on investigator opinion, to a maximum of 30 mg/kg/day GWP42003-P.
  Clobazam (CLB) was administered in line with the physician's preferred CLB dosing regimen for each participant.
  Interventions: Drug: GWP42003-P; Drug: Clobazam

INTERVENTIONS:
Drug: GWP42003-P — GWP42003-P was presented as an oral solution containing 100 mg/milliliter (mL) cannabidiol (CBD) in the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL). Participants received up to a maximum of 30 mg/kg/day.
  Other Names: Cannabidiol (CBD); Epidiolex
Drug: Clobazam — Participants were taking CLB upon entry into the OLE phase of the trial. CLB was not an investigational medicinal product (IMP) for the OLE phase and was not administered by the Sponsor, but was administered at the physician's discretion, as required for each participant. CLB could be stopped, if clinically indicated, without impact on analysis.
  Other Names: CLB

SUMMARY:
This study consisted of 2 parts: a double-blind (DB) phase and an open-label extension (OLE) phase. Only the OLE phase is described in this record. The OLE phase was a safety study. All participants received GWP42003-P initially titrated to 20 milligrams (mg)/kilograms (kg)/day; however, investigators subsequently decreased or increased the participant's dose to a maximum of 30 mg/kg/day (no minimum).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must have had epilepsy, as determined by the investigator, and must have been taking CLB.
* Participant must have had a documented magnetic resonance imaging/computerized tomography of the brain ruling out a progressive neurologic condition.
* Participant must have experienced at least 1 seizure of any type (that is, convulsive: tonic-clonic, tonic, clonic, atonic; focal: focal seizures with retained consciousness and a motor component, focal seizures with impaired consciousness, focal seizures evolving to bilateral secondary generalization) within the 2 months prior to randomization.
* Participant must have been taking CLB and no more than 2 other antiepileptic drugs (AEDs) during the course of the study. However, any participants who were taking these medications after screening were not withdrawn from the study unless there were safety concerns.
* AED(s), including CLB, must have been stable for 4 weeks prior to screening and regimen must have remained stable throughout the duration of the double-blind phase of the study.
* Intervention with vagus nerve stimulation and/or ketogenic diet must have been stable for 4 weeks prior to Baseline and participant/caregiver must have been willing to maintain a stable regimen throughout the double-blind phase of the study.

Key Exclusion Criteria:

* Participant had clinically significant unstable medical conditions other than epilepsy.
* Participants were on CLB at doses above 20 mg per day.
* Participants taking CLB intermittently as rescue medication.
* Participant had a history of symptoms related to a drop in blood pressure due to postural changes (for example, dizziness, light-headedness, blurred vision, palpitations, weakness, syncope).
* Participant had any history of suicidal behavior or any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale in the last month or at screening.
* Participant had clinically relevant symptoms or a clinically significant illness, other than epilepsy in the 4 weeks prior to screening or enrollment, other than epilepsy.
* Participant had consumed alcohol during the 7 days prior to enrollment and was unwilling to abstain during the double-blind phase of the study.
* Participant was currently using or has in the past used recreational or medicinal cannabis, or synthetic cannabinoid-based medications (including Sativex®) within the 3 months prior to study entry.
* Participant had any known or suspected history of any drug abuse or addiction.
* Participant was unwilling to abstain from recreational or medicinal cannabis, or synthetic cannabinoid-based medications (including Sativex) for the duration for the study.
* Participant consumed grapefruit or grapefruit juice 7 days prior to enrollment and was unwilling to abstain from drinking grapefruit juice within 7 days of pharmacokinetic visits.
* Participant had any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP, for example, sesame oil.
* Participant received an IMP within the 12 weeks prior to the screening visit.
* Participant had significantly impaired hepatic function at the screening or randomization visit, defined as any of the following: (A) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN). (B) ALT or AST > 3 × ULN and total bilirubin > 2 × ULN or international normalized ratio > 1.5. (C) ALT or AST > 3 × ULN with the presence of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Barcelona, Spain
- United Kingdom (4):
  - Birmingham
  - Brighton
  - Leeds
  - Salford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled by invitation into the open-label extension (OLE) phase after completing the double-blind phase of the study.
Pre-assignment Details: Two of the 18 participants withdrew during the OLE titration period: 1 met protocol-specified withdrawal criteria; 1 had GWP42003-P withdrawn due to adverse events (AEs) ongoing at entry to the OLE phase.
Groups:
- GWP42003-P: Participants who transferred from the double blind (DB) phase (NCT02565108) to the OLE (still blinded at that stage) tapered off their GWP42003-P or placebo treatment by reducing their maintenance dose by 10% per day and concomitantly titrating GWP42003-P to 20 mg/kg/day initially for the OLE; doses could then be adjusted up or down, dependent on investigator opinion, to a maximum of 30 mg/kg/day GWP42003-P.
  Clobazam (CLB) was administered in line with the physician's preferred CLB dosing regimen for each participant.
Period: Overall Study
Arm/Group | GWP42003-P
Started | 18
Received at Least 1 Dose of Study Drug | 18
Completed OLE Titration Period (OLE population: enrolled participants with ≥1 dose of study drug from Day 2 of Visit 4 onwards.) | 16
Completed | 7
Not Completed | 11
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 1
Not completed — Participant Withdrawn by Investigator | 1
Not completed — Withdrawal by Subject | 1
Not completed — Low Efficacy | 1
Not completed — Participant Met Withdrawal Criteria | 1

BASELINE CHARACTERISTICS:
Population: The study population included all participants who completed the GWEP1428 double-blind phase and entered the OLE phase of the study.
Groups:
- GWP42003-P: Participants who transferred from the DB phase (NCT02565108) to the OLE (still blinded at that stage) tapered off their GWP42003-P or placebo treatment by reducing their maintenance dose by 10% per day and concomitantly titrating GWP42003-P to 20 mg/kg/day initially for the OLE; doses could then be adjusted up or down, dependent on investigator opinion, to a maximum of 30 mg/kg/day GWP42003-P.
  CLB was administered in line with the physician's preferred CLB dosing regimen for each participant.
Arm/Group | GWP42003-P
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.35 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Any History Of Current Seizures [Count of Participants; unit: Participants] | 18

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe OLE-Emergent AEs
Description: An OLE-emergent AE was defined as an AE with an onset date after the first dose of IMP in the OLE phase of the study. The number of participants who experienced 1 or more severe OLE-emergent AEs after the first dose of IMP in the OLE phase of the study up to the Safety follow-up visit (28 [± 3] days following the last dose of IMP) is presented.
  A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Postdose on Day 2 of Visit 4 up to Safety follow-up (28 [± 3] days following the last dose of IMP)
Population: The OLE population included all participants who completed the double-blind phase and entered the OLE phase of the study. The OLE population was the primary analysis set for all safety endpoints reported.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P
Number analyzed (Participants) | 18
Participants | 4

ADVERSE EVENTS:
Time Frame: Postdose on Day 2 of Visit 4 up to Safety follow-up (28 [± 3] days following the last dose of IMP)
Description: The number of participants who experienced OLE-emergent AEs after the first dose of IMP in the OLE phase of the study up to the Safety follow-up visit (28 [± 3] days following the last dose of IMP) is presented. The OLE population was the primary analysis set for all safety endpoints reported. Participants' expected seizure types were not routinely documented as AEs. However, any worsening, including change in the pattern or severity of seizures, was documented as an AE.
Arm/Group | GWP42003-P
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P (N=18)
Alanine aminotransferase abnormal (Investigations) | 1
Aspartate aminotransferase abnormal (Investigations) | 1
Gamma-glutamyltransferase abnormal (Investigations) | 1
Seizure (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P (N=18)
Diarrhoea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Gait disturbance (General disorders) | 1
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 1
Respiratory tract infection (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Eczema infected (Infections and infestations) | 1
Infected bite (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Eosinophil count increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Somnolence (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 4
Seizure (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Irritability (Psychiatric disorders) | 2
Abnormal behaviour (Psychiatric disorders) | 1
Affect lability (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Tearfulness (Psychiatric disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-01-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT02564952/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT02564952/SAP_001.pdf